CLINICAL TRIAL: NCT01622517
Title: Computed Tomography Perfusion (CTP) to Predict Response to Recanalization in Ischemic Stroke Project
Brief Title: Computed Tomography Perfusion (CTP) to Predict Response to Recanalization in Ischemic Stroke Project (CRISP)
Acronym: CRISP
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Saint Luke's Health System (Other); University of Pittsburgh (Other); Emory University (Other); Chatanooga Center for Neurological Research (Unknown); University of Miami (Other)
Responsible Party: Principal Investigator, Maarten Lansberg, Assistant Professor, Stanford University
Other Study IDs: 22227
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall goal of the CTP to predict Response to recanalization in Ischemic Stroke Project (CRISP) is to develop a practical tool to identify acute stroke patients who are likely to benefit from endovascular therapy.

The project has two main parts. During the first part, the investigators propose to develop a fully automated system (RAPID) for processing of CT Perfusion (CTP) images that will generate brain maps of the ischemic core and penumbra. There will be no patient enrollment in part one of this project.

During the second part, the investigators aim to demonstrate that physicians in the emergency setting, with the aid of a fully automated CTP analysis program (RAPID), can accurately predict response to recanalization in stroke patients undergoing revascularization. To achieve this aim the investigators will conduct a prospective cohort study of 240 consecutive stroke patients who will undergo a CTP scan prior to endovascular therapy. The study will be conducted at four sites (Stanford University, St Luke's Hospital, University of Pittsburgh Medical Center, and Emory University/Grady Hospital). Patients will have an early follow-up MRI scan within 12+/-6 hours to assess reperfusion and a late follow-up MRI scan at day 5 to determine the final infarct.

ELIGIBILITY:
Inclusion Criteria:

1. be 18 or older;
2. have a clinical diagnosis of ischemic stroke and a score of 5 or more points on the NIHSSS;
3. be scheduled to undergo intraarterial (IA) therapy for acute hemispheric stroke (either as primary therapy or as adjuvant therapy following intravenous tPA treatment);
4. be scheduled to have a standard CT including perfusion imaging and CT angiography of the circle of Willis (CTA) prior to IA therapy;
5. begin intra-arterial thrombectomy within 90 minutes of completion of the CT scan and within 18 hours of symptom onset. (Start of IA therapy is defined as the time of insertion of the femoral artery sheath; Time of brain scan is defined as the time that the scan is completed); and
6. have provided informed consent.

Exclusion Criteria:

1. have any pre-existing illness resulting in a modified Rankin Scale Score of 3 or higher prior to the qualifying stroke;
2. are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
NIHSS Score | 30 Day
  A "favorable clinical response", defined as an 8-point or more improvement on the NIH score when comparing the baseline score to the 30-day score or a 30-day NIH score of 0-1, will be the primary endpoint for the study

SECONDARY OUTCOMES:
modified Rankin Score | 90 day
  90 day modified Rankin Score 0-2, 90 day modified Rankin distribution, and 90 day Rankin Score 0-1

CONTACTS AND LOCATIONS:
Overall Officials: Maarten G Lansberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

REFERENCES:
- [Derived] Dehkharghani S, Lansberg M, Venkatsubramanian C, Cereda C, Lima F, Coelho H, Rocha F, Qureshi A, Haerian H, Mont'Alverne F, Copeland K, Heit J. High-Performance Automated Anterior Circulation CT Angiographic Clot Detection in Acute Stroke: A Multireader Comparison. Radiology. 2021 Mar;298(3):665-670. doi: 10.1148/radiol.2021202734. Epub 2021 Jan 12. PMID 33434110